CLINICAL TRIAL: NCT02242435
Title: A Randomized, Placebo-controlled, Double-blind Study to Evaluate the Safety and Efficacy of Three Intra-articular Injections of Ampion™ (4 mL) Administered Two Weeks Apart in Adults With Pain Due to Osteoarthritis of the Knee
Brief Title: A Multiple Injection Study Evaluating Safety and Efficacy of Ampion in Osteoarthritis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Ampio Pharmaceuticals. Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: AP-008
Record Dates: First submitted 2014-09-15; First posted 2014-09-17 (Estimated); Results first posted 2022-08-29 (Actual); Last update posted 2022-09-15 (Actual); Status verified 2022-08

CONDITIONS: Osteoarthritis of the Knee
Keywords: Osteoarthritis; osteoarthritis of the knee
MeSH Terms: conditions — Osteoarthritis, Knee; Osteoarthritis | interventions — Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Ampion 4ml dose (Experimental): 4 mL intra-articular injection of Ampion
  Interventions: Biological: 4 mL injection of Ampion
- Placebo Solution (Placebo Comparator): 4 mL placebo intra-articular injection
  Interventions: Drug: 4 mL Injection of Placebo

INTERVENTIONS:
Biological: 4 mL injection of Ampion — 4 mL injection of Ampion
  Arms: Ampion 4ml dose
Drug: 4 mL Injection of Placebo
  Other Names: Saline
  Arms: Placebo Solution

SUMMARY:
This study will evaluate the efficacy of three intra-articular injections, given 2 weeks apart, of Ampion™ in Adults with pain due to osteoarthritis of the knee.

DETAILED DESCRIPTION:
A randomized, placebo-controlled, double-blinded study to evaluate the efficacy and safety of repeated intra-articular injections of Ampion™ in adult subjects with advanced osteoarthritis of the knee.

The primary study objective was to evaluate the efficacy and safety from Baseline to Week 20 of 3 Ampion™ 4 mL intra-articular (IA) injections vs saline administered 2 weeks apart in improving knee pain in subjects suffering from osteoarthritis (OA) of the knee (OAK).

The secondary study objective was to analyze the effect of Ampion 4 mL vs saline on a change in Patient's Global Assessment (PGA) and knee function from Baseline to Week 20.

ELIGIBILITY:
Inclusion Criteria:

1. Able to provide written informed consent to participate in the study.
2. Willing and able to comply with all study requirements and instructions of the site study staff.
3. Male or female, 40 years to 85 years old (inclusive).
4. Must be ambulatory.
5. Index knee must be symptomatic for greater than 6 months with a clinical diagnosis of OA and supported by radiological evidence (x-ray) acquired at screening and assessed by a central reader. Subjects must have a Kellgren Lawrence Grade of III or IV for inclusion in the study.
6. Moderate to moderately-severe OA pain in the index knee (rating of at least 1.5 on the WOMAC® Index 3.1 5-point Likert Pain Subscale) assessed at screening and confirmed at randomization.
7. Moderate to moderately-severe OA pain in the index knee (even if chronic doses of non-steroidal anti-inflammatory drug [NSAID], which have not changed in the 4 weeks prior to screening, have been/are being used).
8. No analgesia taken 24 hours before efficacy measure.

Exclusion Criteria:

1. As a result of medical review and screening investigation, the Principal Investigator considers the subject unfit for the study.
2. Previous Ampion™ injection in the index knee.
3. Known clinically significant liver abnormality (e.g., cirrhosis, transplant, etc).
4. A history of allergic reactions to human albumin (reaction to non-human albumin such as egg albumin is not an exclusion criterion).
5. A history of allergic reactions to excipients in 5% human albumin (N-acetyltryptophan, sodium caprylate).
6. Presence of tense effusions in the index knee.
7. Inflammatory or crystal arthropathies, acute fractures, history of aseptic necrosis or joint replacement in the index knee, as assessed locally by the Principal Investigator.
8. Isolated patella femoral syndrome, also known as chondromalacia, in the index knee.
9. Any other disease or condition interfering with the free use and evaluation of the index knee for the duration of the trial (e.g., cancer, congenital defects, spine OA).
10. Major injury to the index knee within the 12 months prior to screening.
11. Severe hip OA ipsilateral to the index knee.
12. Any pain that could interfere with the assessment of index knee pain (e.g., pain in any other part of the lower extremities, pain radiating to the knee).
13. Any pharmacological or non-pharmacological treatment targeting OA started or changed during the 4 weeks prior to treatment or likely to be changed during the duration of the study.
14. Use of the following medications are exclusionary:

    1. IA injected pain medications in the study knee during the study;
    2. Analgesics containing opioids. NSAIDs may be continued at levels preceding the study and acetaminophen is available as a rescue medication during the study from the provided supply;
    3. Topical treatment on osteoarthritis index knee during the study;
    4. Significant anticoagulant therapy (e.g., Heparin or Lovenox) during the study (treatment such as Aspirin and Plavix are allowed);
    5. Systemic treatments that may interfere with safety or efficacy assessments during the study;
    6. Immunosuppressants;
    7. Use of corticosteroids > 10 mg prednisolone equivalent per day (if ≤ 10 mg prednisolone, the dose must be stable).
15. Any human albumin treatment in the 3 months before randomization.

Ages: 40 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 342 (Actual)
Dates: Start 2014-09 (Actual); Primary Completion 2015-04 (Actual); Study Completion 2015-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Howard Levy, M.D., Study Director — Ampio Pharmaceuticals. Inc.
Locations (1):
- Ampio Pharmaceuticals, Inc., Englewood, Colorado, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment of subjects occurred in medical clinics during the months of September, October, and November 2014.
Pre-assignment Details: No pharmacological or non-pharmacological treatment targeting osteoarthritis (OA) started or changed during the 4 weeks prior to randomization or likely to be changed during the duration of the study.
Groups:
- Ampion 4 mL: 4 mL intra-articular injection of Ampion
  Ampion <5 kilodalton (kDa) ultrafiltrate of 5% human serum albumin: 4 mL intra-articular injection of Ampion
- Placebo 4 mL: 4 mL placebo intra-articular injection
  Placebo: Saline
Period: Overall Study
Arm/Group | Ampion 4 mL | Placebo 4 mL
Started | 172 | 170
Completed | 152 | 154
Not Completed | 20 | 16
Not completed — Lost to Follow-up | 3 | 4
Not completed — Adverse Event | 3 | 2
Not completed — Withdrawal by Subject | 13 | 8
Not completed — Death | 0 | 1
Not completed — Protocol Violation | 1 | 0
Not completed — Physician Decision | 0 | 1

BASELINE CHARACTERISTICS:
Population: Intent to Treat (ITT)
Groups:
- Ampion 4 mL: 4 mL intra-articular injection of Ampion
  Ampion <5 kDa ultrafiltrate of 5% human serum albumin
- Total: Total of all reporting groups
Arm/Group | Ampion 4 mL | Placebo 4 mL | Total
Number analyzed (Participants) | 172 | 170 | 342
Age, Continuous [Mean (Standard Deviation); unit: years] | 63.3 (9.1) | 63.2 (9.5) | 63.2 (9.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 93 | 105 | 198
  Male | 79 | 65 | 144
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 11 | 12 | 23
  Not Hispanic or Latino | 161 | 158 | 319
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 1
  Asian | 1 | 1 | 2
  Native Hawaiian or Other Pacific Islander | 1 | 2 | 3
  Black or African American | 22 | 36 | 58
  White | 146 | 130 | 276
  More than one race | 1 | 1 | 2
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 172 | 170 | 342
Weight (kg) [Mean (Standard Deviation); unit: kg] | 96.2 (23.8) | 96.4 (22.5) | 96.3 (23.2)
BMI (kg/m^2) [Mean (Standard Deviation); unit: kg/m^2] | 34.3 (7.5) | 34.9 (8.0) | 34.6 (7.8)
Kellgren-Lawrence (KL) Grade [Count of Participants; unit: Participants] — Kellgren-Lawrence grading is based on the radiologic features of osteoarthritis.
  Ann Rheum Dis. 1957;16:494-502.
  Grade III (Moderate): Moderate osteophytes, definite joint space narrowing, some sclerosis, possible bone-end deformity.
  Grade IV (Severe): Large osteophytes, marked joint space narrowing, severe sclerosis, definite bone ends deformity.
  Participants
    Kellgren-Lawrence Grade III | 50 | 64 | 114
    Kellgren-Lawrence Grade IV | 122 | 106 | 228
WOMAC Pain [Mean (Standard Deviation); unit: score on a scale] — The Western Ontario and McMaster Universities Arthritis Index (WOMAC) 3.1 evaluates Pain (5 items): during walking, using stairs, in bed, sitting or lying, and standing upright.
  Subjects respond to each subscale by using a 5-point Likert score. (0=none; 1=mild; 2=moderate; 3=severe; 4=extreme). Mean of the 5 scores constitutes the Baseline Pain Score.
  The minimum score on this scale is 0, and the maximum score is 4. Higher scores are indicative of higher levels of self-reported pain.
  score on a scale | 2.51 (0.57) | 2.57 (0.61) | 2.54 (0.59)
WOMAC Function [Mean (Standard Deviation); unit: score on a scale] — WOMAC 3.1 evaluates Physical Function (17 items): using stairs, rising from sitting, standing, bending, walking, getting in/out of a car, shopping, putting on/taking off socks, rising from bed, lying in bed, getting in/out of bath, sitting, getting on/off toilet, heavy/light domestic duties.
  Subjects respond to each by using a 5-point Likert score. (0=none; 1=mild; 2=moderate; 3=severe; 4=extreme). Mean of the 17 scores constitutes the Baseline Function Score. Minimum score is 0; maximum is 4.
  Higher scores indicate of higher levels of limitations of self-reported physical function.
  score on a scale | 2.51 (0.63) | 2.59 (0.61) | 2.55 (0.62)

OUTCOME MEASURES:

1. Primary Outcome: Change in Knee Pain
Description: Mean Change in WOMAC A Pain (Western Ontario and McMaster Universities Arthritis Index) score from Baseline to 12 weeks. 5-point Likert scale (0=none to 4=extreme). A negative difference constitutes a decrease in pain with a greater negative value indicating a greater reduction in pain.
Time Frame: Scored at Baseline and 20 Weeks
Population: Intent to Treat (ITT)
Measure: Mean (95% Confidence Interval); unit: score on a scale
Groups:
- Ampion 4 mL Injection: 4 mL intra-articular injection of Ampion
  Ampion: <5 kDa ultrafiltrate of 5% human serum albumin
- Placebo 4 mL Injection: 4 mL placebo intra-articular injection
  Placebo: Saline
Arm/Group | Ampion 4 mL Injection | Placebo 4 mL Injection
Number analyzed (Participants) | 172 | 170
score on a scale | -0.96 [-1.09 to -0.82] | -1.10 [-1.24 to -0.95]
Statistical Analysis 1: Comparison: Ampion 4 mL Injection vs Placebo 4 mL Injection; Test type: Superiority; p = 0.26, ANCOVA — Adjusted for baseline WOMAC score

2. Secondary Outcome: Change in Knee Function
Description: Mean change in WOMAC C function score (Western Ontario and McMaster Universities Arthritis Index) from Baseline to 12 weeks. 5-point Likert scale indicating limitation of function (0=none to 4=extreme). A greater negative value indicates a improvement in function.
Time Frame: Scored at Baseline and 20 Weeks
Population: Intent to Treat (ITT)
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Ampion 4 mL Injection | Placebo 4 mL Injection
Number analyzed (Participants) | 172 | 170
score on a scale | -0.94 [-1.08 to -0.81] | -1.08 [-1.22 to -0.94]
Statistical Analysis 1: Comparison: Ampion 4 mL Injection vs Placebo 4 mL Injection; Test type: Superiority; p = 0.30, ANCOVA — Adjustment for baseline WOMAC score

ADVERSE EVENTS:
Time Frame: 24 Weeks
Description: Patients will be followed for the occurrence of Adverse Events (AEs) from Baseline through Week 24.
Groups:
- Ampion 4 mL: 4 mL intra-articular injection of Ampion
  Ampion <5 kDa ultrafiltrate of 5% human serum albumin: 4 mL intra-articular injection of Ampion
Arm/Group | Ampion 4 mL | Placebo 4 mL
All-Cause Mortality (participants affected / at risk) | 0/172 | 1/170
Serious Adverse Events (participants affected / at risk) | 4/172 | 11/170
Other Adverse Events (participants affected / at risk) | 107/172 | 125/170
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Ampion 4 mL (N=172) | Placebo 4 mL (N=170)
Plasma Cell Myeloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2
Salivary Gland Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Incisional Hernia (Injury, poisoning and procedural complications) | 1 | 0
Injury (Injury, poisoning and procedural complications) | 0 | 1
Joint Injury (Injury, poisoning and procedural complications) | 0 | 1
Abcess Limb (Infections and infestations) | 0 | 1
Gastroenteritis (Infections and infestations) | 0 | 1
Influenza (Infections and infestations) | 0 | 1
Transient Ischaemic Attack (Nervous system disorders) | 2 | 0
Angina Unstable (Cardiac disorders) | 0 | 1
Atrial Fibrillation (Cardiac disorders) | 1 | 0
Angioedema (Skin and subcutaneous tissue disorders) | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Ampion 4 mL (N=172) | Placebo 4 mL (N=170)
Nausea (Gastrointestinal disorders) | 0 | 4
Injection Site Bruising (General disorders) | 3 | 3
Injection Site Pain (General disorders) | 11 | 10
Injection Site Swelling (General disorders) | 2 | 3
Oedema Peripheral (General disorders) | 1 | 4
Pain (General disorders) | 3 | 0
Bronchitis (Infections and infestations) | 5 | 6
Gastroenteritis (Infections and infestations) | 3 | 4
Influenza (Infections and infestations) | 1 | 3
Nasopharyngitis (Infections and infestations) | 5 | 1
Respiratory Tract Infection Viral (Infections and infestations) | 3 | 0
Sinusitis (Infections and infestations) | 5 | 4
Upper Respiratory Tract Infection (Infections and infestations) | 10 | 10
Contusion (Injury, poisoning and procedural complications) | 7 | 4
Fall (Injury, poisoning and procedural complications) | 2 | 4
Joint Injury (Injury, poisoning and procedural complications) | 4 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 19 | 21
Back Pain (Musculoskeletal and connective tissue disorders) | 0 | 4
Joint Stiffness (Musculoskeletal and connective tissue disorders) | 4 | 4
Joint Swelling (Musculoskeletal and connective tissue disorders) | 3 | 6
Pain in Extremity (Musculoskeletal and connective tissue disorders) | 3 | 4
Plantar Fasciitis (Musculoskeletal and connective tissue disorders) | 1 | 3
Headache (Nervous system disorders) | 5 | 3
Cough (Respiratory, thoracic and mediastinal disorders) | 3 | 2
Hypertension (Vascular disorders) | 3 | 8
Bursitis (Musculoskeletal and connective tissue disorders) | 0 | 3
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 | 3
Rash (Skin and subcutaneous tissue disorders) | 1 | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less